CLINICAL TRIAL: NCT00425113
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of Metronidazole Combined With Antituberculous Chemotherapy vs. Antituberculous Chemotherapy With Placebo in Subjects With Multi-Drug Resistant Pulmonary Tuberculosis
Brief Title: Metronidazole for Pulmonary Tuberculosis (South Korea)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 999907041; 07-I-N041
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-05

CONDITIONS: Tuberculosis; Multi-Drug Resistant Tuberculosis
Keywords: Mycobacterium Tuberculosis; Anaerobic; FDG-PET-HRCT; HRCT; Lesion Matrix; Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant | interventions — Metronidazole; Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Experimental): Metronidazole added to background TB treatment regimen during initial 2 months
  Interventions: Drug: Metronidazole; Procedure: Blood Draw; Procedure: CT Scan; Procedure: PET Scan
- Placebo (Placebo Comparator): Placebo added to background TB treatment regimen during initial 2 months
  Interventions: Procedure: Blood Draw; Procedure: CT Scan; Procedure: PET Scan

INTERVENTIONS:
Drug: Metronidazole
  Arms: Metronidazole
Procedure: Blood Draw
Procedure: CT Scan
Procedure: PET Scan

SUMMARY:
This study will evaluate the effect of adding metronidazole to standard second-line therapy for tuberculosis in patients who have multi-drug resistant tuberculosis (MDR-TB) of the lungs. It will evaluate the safety and tolerability of metronidazole in combination with antituberculosis agents. Metronidazole is a drug widely used to treat bacterial and parasitic infections occurring in environments with very little oxygen such as the human colon. Nine million new cases of sputum-positive tuberculosis are diagnosed worldwide each year.

Patients ages 20 and older who have symptoms of TB, who have been treated for tuberculosis but whose disease is multi-drug resistant, and who are not pregnant or breast feeding may be eligible for this study. They will be recruited in the National Masan Tuberculosis Hospital (NMTH), Masan, Republic of Korea. Patients will undergo the following tests and procedures:

* Collection of sputum for counting of bacteria.
* Drawing of blood for routine blood chemistry analysis; for measuring levels of metronidazole; TB lipid analysis; and for testing levels of T-cells, which are part of an immune response.
* Two targeted positron emission tomography (PET) scans, each with a computed tomography (CT) scan, and five high-resolution CT scans.

Patients will receive either an 8-week course of standard second-line agents plus placebo (sugar pill) or an 8-week course of standard agents plus metronidazole. The subjects, doctors and researchers will not know which patients are taking the metronidazole until after the first 2 years of the trial. A total of 60 patients will be assigned to two cohorts of 30 patients each. After 8 weeks, all patients will return to the standard of care chemotherapy, according to normal procedures at NMTH.

Side effects of metronidazole commonly reported are vaginal discharge, symptoms of Candida cervicitis and vaginitis, headache, nausea and vomiting, and dizziness. Peripheral neuropathy, an abnormal condition of the nerves, may also be a side effect. The precise incidence of neuropathy is unknown but is usually related to the duration of metronidazole use. It can almost always be reversed when the drug is discontinued. Serious side effects, though rare, may include leukopenia and thrombocytopenia (disorders in the blood), seizures and other central nervous system problems, and hepatitis.

This study may or may not have a direct benefit for participants. However, it is possible that patients' drug-resistant disease may be more effectively treated as a result of metronidazole. The study may help identify new methods for measuring drug effectiveness during TB studies.

DETAILED DESCRIPTION:
BACKGROUND:

Despite significant in vitro data that metronidazole is active against Mycobacterium tuberculosis (MTB) maintained under anaerobic conditions, the utility of this agent has not been evaluated carefully in human disease due to lack of efficacy in murine models of tuberculosis (TB). Unlike disease in rodents, however, human disease is characterized by discrete types of lesions including both aerobic (cavities) and anaerobic (caseous necrotic nodules) areas. Recent experiments in non-human primates have demonstrated that closed caseous necrotic lesions are highly anoxic and are, therefore, likely to contain anaerobic bacilli highly susceptible to metronidazole. Recent studies in TB-infected rabbits have shown that metronidazole therapy is highly effective in an animal model that recapitulates this feature of human disease. Both of these studies support the possibility that metronidazole may have unique activity against an anaerobic sub-population of bacilli in human disease. Such sub-populations may be responsible for the extended duration of chemotherapy typically employed in tuberculosis chemotherapy, as anoxic bacteria are highly resistant to the sterilizing effects of front-line tuberculosis agents. One small clinical trial of metronidazole in an Indian population also suggests that this agent may have a significant unappreciated role in the control of human tuberculosis.

AIMS:

The major aim of this study is to evaluate the ability of metronidazole to kill an anaerobic sub-population of Mycobacterium tuberculosis within multi-drug resistant tuberculosis (MDR-TB) patients. In order to address this sub-population in the context of disease, this study combines traditional measurements of drug efficacy, including the rate of sputum clearance of organisms, with a functional imaging technique, [(18) F]-fluoro-2-deoxy-D-glucose -positron emission tomography - high-resolution computed tomography (FDG-PET-HRCT) that has not previously been applied to monitoring tuberculosis chemotherapy. In addition, this clinical trial will evaluate the tolerability and preliminary efficacy of metronidazole (500 mg three times a day (t.i.d.) when given in combination with standard second-line antituberculous treatment.

METHODS:

Type of study to be conducted:

Randomized, double-blinded, placebo controlled phase II study.

Population to be Studied:

The study population will be drawn from subjects at the National Masan Tuberculosis Hospital (NMTH), Changwon, Republic of Korea. Subjects presenting at NMTH who have been previously treated with first-line agents and who are multi-drug resistant (MDR), defined as having TB isolates that are resistant to at least isoniazid and rifampicin, and are therefore eligible for second-line antituberculous drug therapy will be included.

Treatment Regimen and Treatment Period(s):

All patients will receive either: (1) an 8-week course of standard second-line agents plus placebo t.i.d., or (2) an 8-week course of standard second-line agents plus 500 mg t.i.d. metronidazole. In total, sixty subjects will be accrued into two cohorts of 30 patients each. After 8 weeks, all subjects will revert to standard of care (SOC) chemotherapy according to normal procedures at NMTH. According to hospital standard of care, patients are continued on second-line medications for 18-24 months following sputum culture conversion.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and females age 20 and above
  2. Signs or symptoms of tuberculosis (i.e., cough that has lasted 3 weeks or longer, hemoptysis, chest pain, fatigue, weight loss, night sweats)
  3. Subjects with documented AFB smear-positive pulmonary tuberculosis at screening to NMTH
  4. Radiographic evidence of tuberculous disease of the lung(s)
  5. TB isolate resistant to at least isoniazid and rifampicin
  6. Drug Susceptibility Testing (DST) results known for ofloxacin (can be either sensitive or resistant)
  7. Ability and willingness to give written or oral informed consent
  8. Willingness to be an inpatient at NMTH for, at minimum, the duration of study drug/placebo treatment
  9. Willingness to have samples stored
  10. Available for follow-up visits

EXCLUSION CRITERIA:

1. People who are unwilling or unable to abstain from alcohol consumption for the study drug treatment duration (8 weeks)
2. Women of childbearing potential, who are pregnant, breast feeding, or unwilling to avoid pregnancy by the use of appropriate contraception including oral and subcutaneous implantable hormonal contraceptives, condoms, diaphragm, intrauterine device (IUD), or abstinence from sexual intercourse at study screening and during the study drug/placebo treatment (two months with allowed stops) (Note: Prospective female participants of childbearing potential must have negative pregnancy test (urine) within 48 hours prior to study entry.)
3. Subjects with pan resistant isolates
4. Presently taking 2nd -line agents started more than 14 days prior to initial FDG-PET scan
5. People with any of the following in their current medical assessment:

   1. Absolute neutrophil count less than 1000 cells/mL
   2. White Blood Cell count (WBC) less than 3.0 X 10(3)/microliter
   3. Hemoglobin less than 7.0 g/dL
   4. Platelet count less than 75,000 cells/mm(3)
   5. Serum creatinine greater than 2.0 mg/dL
   6. Aspartate aminotransferase (AST or SGOT) greater than 100 IU/L
   7. Alanine aminotransferase (ALT or SGPT) greater than 100 IU/L
   8. Total bilirubin greater than 2 mg/dL
   9. Moderate or severe peripheral neuropathy
   10. HIV-1 or HIV-2 infection
   11. History of systemic lupus erythematosus, rheumatoid arthritis, or other connective tissue disease
6. Terminal illness with impending mortality
7. History of allergy or serious adverse reaction to metronidazole or placebo formulation used in this study
8. The use of any of the following drugs within 30 days prior to study or anticipated use of these drugs within the next 60 days:

   1. Systemic cancer chemotherapy
   2. Systemic corticosteroids
   3. Systemic investigational agents
   4. Antiretroviral medications
   5. Growth factors
   6. HIV vaccines
   7. Immune globulin
   8. Interleukins
   9. Interferons
9. The need for ongoing therapy with warfarin, phenytoin, lithium, cimetidine, disulfiram, ergot derivatives, cholestyramine, fosphenytoin, carbamazepine, cyclosporine, tacrolimus, sirolimus, amiodarone or phenobarbital while on study drug.
10. Any other serious systemic illness requiring treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy for at least 14 days prior to study entry
11. Unwilling to be an inpatient at NMTH for greater than or equal to 2 months
12. Any condition that the investigator believes would warrant exclusion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-12; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- South Korea (2):
  - National Masan Tuberculosis Hospital, Masan
  - Yonsei University College of Medicine, Seoul

REFERENCES:
- [Background] Andreu J, Caceres J, Pallisa E, Martinez-Rodriguez M. Radiological manifestations of pulmonary tuberculosis. Eur J Radiol. 2004 Aug;51(2):139-49. doi: 10.1016/j.ejrad.2004.03.009. PMID 15246519
- [Background] Brooks JV, Furney SK, Orme IM. Metronidazole therapy in mice infected with tuberculosis. Antimicrob Agents Chemother. 1999 May;43(5):1285-8. doi: 10.1128/AAC.43.5.1285. PMID 10223954
- [Background] Carrara S, Vincenti D, Petrosillo N, Amicosante M, Girardi E, Goletti D. Use of a T cell-based assay for monitoring efficacy of antituberculosis therapy. Clin Infect Dis. 2004 Mar 1;38(5):754-6. doi: 10.1086/381754. Epub 2004 Feb 17. PMID 14986262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pulmonary multidrug-resistant tuberculosis subjects were recruited from the National Masan Hospital, Masan, South Korea from 2009-2010.
Groups:
- Metronidazole: Subjects were randomized to receive metronidazole 500 mg TID or placebo for 8 weeks, in addition to an individualized background TB treatment regimen. Total duration of treatment was about 18 months following sputum culture conversion.
Period: Overall Study
Arm/Group | Metronidazole | Placebo
Started | 17 | 18
Exposed to Study Drug | 16 | 17
Completed | 15 (Included in modified intent-to-treat analysis) | 16 (Included in modified intent-to-treat analysis)
Not Completed | 2 | 2
Not completed — uncontrolled diabetes mellitus | 1 | 0
Not completed — diagnosis of abdominal TB | 0 | 1
Not completed — missing study drug more than 14 days | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 2 subjects excluded: 1 for uncontrolled diabetes mellitus and 1 for diagnosis of extrapulmonary TB. 2 additional subjects withdrew: 1 self- withdrew and the other was withdrawn for missing >14 days of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age Continuous [Median (Inter-Quartile Range); unit: years] | 36 [28 to 39] | 38 [31 to 44] | 37 [30 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Changes in TB Lesion Sizes Using High Resolution Computed Tomography (HRCT).
Description: Lesions were defined as nodules (<2 mm, 2-<4 mm, and 4-10 mm), consolidations, collapse, cavities, fibrosis, bronchial thickening, tree-in-bud opacities, and ground glass opacities. Each CT was divided into six zones (upper, middle, and lower zones of the right and left lungs) and independently scored for the above lesions by three separate radiologists blinded to treatment arm. A fourth radiologist adjudicated any scores that were widely discrepant among the initial three radiologists. The HRCT score was determined by visually estimating the extent of the above lesions in each lung zone as follows: 0=0% involvement; 1= 1-25% involvement; 2=26-50% involvement; 3=51-75% involvement; and 4=76-100% involvement. A composite score for each lesion was calculated by adding the score for each specific abnormality in the 6 lung zones and dividing by 6, with the change in composite score measured at 2 and 6 months compared to baseline. Composite sums of all 10 composite scores are reported.
Time Frame: 6 months.
Measure: Mean (Standard Error); unit: reader score
Groups:
- Metronidazole: Subjects were randomized to receive metronidazole 500 mg three times daily or placebo for 8 weeks, in addition to an individualized background TB treatment regimen. Total duration of treatment was about 18 months following sputum culture conversion.
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 15 | 16
reader score
  Baseline composite sum of all 10 features | 8.11 (1.27) | 10.08 (1.00)
  Month 6 composite sum of all 10 features | 6.64 (1.01) | 7.24 (0.89)

2. Secondary Outcome: Time to Sputum Culture Conversion to Negative on Solid Medium
Time Frame: 2 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 15 | 16
days | 21 [16 to 71] | 42.5 [15 to 69]

ADVERSE EVENTS:
Arm/Group | Metronidazole | Placebo
Serious Adverse Events (participants affected / at risk) | 9/15 | 4/16
Other Adverse Events (participants affected / at risk) | 11/15 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (N=15) | Placebo (N=16)
peripheral neuropathy (Nervous system disorders) | 4 (4) | 0 (0)
hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
seizure (Nervous system disorders) | 3 (3) | 1 (1)
aspergilloma (Infections and infestations) | 1 (1) | 0 (0)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (N=15) | Placebo (N=16)
hyperuricemia (General disorders) | 6 (7) | 6 (6)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
peripheral neuropathy (Nervous system disorders) | 4 (4) | 2 (2)
hyperglycemia (Endocrine disorders) | 2 (2) | 2 (2)
hypokalemia (General disorders) | 1 (1) | 0 (0)
hypercholesterolemia (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Major limitation of our study was the small sample size. Planned enrollment was 80 subjects but DSMB recommended closing the study to new enrollment after 35 subjects due to increased peripheral neuropathy in the metronidazole arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes